CLINICAL TRIAL: NCT00017459
Title: The International Tirazone Triple Trial (i3T): A Phase III, Randomized Efficacy And Safety Study Of The Combination Chemotherapy With Tirapazamine+Cisplatin+Vinorelbine Versus Cisplatin+Vinorelbine In Subjects With Inoperable, Previously Untreated, Non-Small Cell Lung Cancer
Brief Title: Cisplatin Plus Vinorelbine With or Without Tirapazamine in Treating Patients With Stage IIIB or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SANOFI-EFC3675; CDR0000068690 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-06-06; First posted 2004-02-16 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Tirapazamine; Vinorelbine

INTERVENTIONS:
Drug: cisplatin
Drug: tirapazamine
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if cisplatin and vinorelbine are more effective with or without tirapazamine in treating non-small cell lung cancer

PURPOSE: Randomized phase III trial to compare the effectiveness of cisplatin plus vinorelbine with or without tirapazamine in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the overall survival duration of patients with stage IIIB or IV non-small cell lung cancer treated with vinorelbine and cisplatin with or without tirapazamine. II. Compare the complete and partial response rates, time to disease progression, and time to treatment failure in these patients treated with these regimens. III. Compare the clinical benefit of these regimens, in terms of performance status and body weight, in these patients. IV. Compare the toxicity and safety of these regimens in these patients. V. Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms. Arm I: Patients receive tirapazamine IV over 2 hours followed by cisplatin IV over 1 hour on day 1. Patients also receive vinorelbine IV over 6-10 minutes on days 1, 8, 15, and 22. Arm II: Patients receive cisplatin and vinorelbine as in arm I. Treatment repeats every 28 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, during each course of treatment, at 30 days after the last course of treatment, and then every 8 weeks for 2-3 years. Patients are followed every 8 weeks for 2-3 years.

PROJECTED ACCRUAL: Approximately 800 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer (NSCLC) Stage IIIB or IV Newly diagnosed or recurrent disease Measurable lesions At least 10 mm by spiral CT scan OR At least 20 mm by conventional techniques Previously irradiated lesions are considered measurable provided they progressed or appeared after completion of radiotherapy The following are considered nonmeasurable: Pleural or pericardial effusions Cystic lesions Lymphangitis pulmonis Bony x-ray abnormalities Abnormal scans with nonmeasurable filling defects No symptomatic brain metastasis or CNS involvement by CT scan or MRI

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine normal Other: No other malignancy within the past 5 years except adequately treated carcinoma in situ of the cervix or basal cell carcinoma that is not likely to recur No history of allergic reactions to diuretics or antiemetics (e.g., 5-HT3 antagonists) used on this study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy or biologic therapy for NSCLC Chemotherapy: No prior chemotherapy for NSCLC No prior platinum-based chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to potential indicator lesion(s) At least 4 weeks since prior radiotherapy and recovered Surgery: Recovered from prior surgical procedure(s) Other: At least 30 days since prior investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-07; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elwyn Y. Loh, MD, Study Chair — Sanofi
Locations (42):
- United States (42):
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Medical Oncology Internal Medicine, Los Angeles, California
  - Bay Area Tumor Institute, Oakland, California
  - Medical Oncology Care Associates, Orange, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Los Angeles County Harbor-UCLA Medical Center, Torrance, California
  - Medical Oncology-Hematology Consultants, P.A., Wilmington, Delaware
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center - Washington, DC, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Watson Clinic, Lakeland, Florida
  - Ocala Research Institute, Inc, Ocala, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Dreyer Medical Clinic, Aurora, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Northwest Oncology and Hematology, S.C., Elk Grove Village, Illinois
  - Rockford Clinic, Rockford, Illinois
  - Cancer Care Center, New Albany, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Hematology-Oncology Clinic, Baton Rouge, Louisiana
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - Capitol Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Western Montana Clinic, Missoula, Montana
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - New York Medical College, Valhalla, New York
  - Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - North Penn Hospital, Lansdale, Pennsylvania
  - Fox Chase - Temple Cancer Center, Philadelphia, Pennsylvania
  - Lone Star Oncology, Austin, Texas
  - Center for Oncology Research and Treatment, Medical City Hospital, Dallas, Texas
  - Southwest Cancer Center at University Medical Center, Lubbock, Texas
  - Baptist Health System Cancer Program, San Antonio, Texas
  - Cancer Therapy Research Center, San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - Arlington-Fairfax Hematology/Oncology, PC, Arlington, Virginia